CLINICAL TRIAL: NCT04011774
Title: PLANning Your Every Day Life I Virtual REality : a Study Schizophrenia. Mathurin Serious Game
Brief Title: Planning Your Everyday Life in Virtual Reality : a Study in Schizophrenia;
Acronym: PlaniRev
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D17-P025
Record Dates: First submitted 2019-04-29; First posted 2019-07-08 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLANI-REV (Experimental): Persons with schizophrenia who will benefit from the fifteen weekly sessions of PLANI-REV group program
  Interventions: Other: PLANI-REV
- RELAXATION (Active Comparator): Persons with schizophrenia who will benefit from a non cognitive stimulation, namely RELAXATION, in a day-care clinic or day-care therapeutic activities center during fifteen weekly sessions. This activity will be 15 groups sessions of relaxation.
  Interventions: Other: RELAXATION

INTERVENTIONS:
Other: PLANI-REV — Cognitive remediation program.
  Arms: PLANI-REV
Other: RELAXATION — Stimulation with no cognitive remediation.
  Arms: RELAXATION

SUMMARY:
Patients with schizophrenia , who visit frenquently day-care or day-care activities clinics, often experience difficulties of daily living and cognitive deficits. Living independently is a key for recovery. Cognitive remediation is a therapy which reduces deficit and improves daily living. Nowadays no program exists targeting neurocognitive functions in virtual reality which could mimic everyday life in a virtual town.

Hypotheses :

* Persons with schizophrenia experience difficulties in daily living and disabilities to plan in everyday life. PLANI-REV program, a serious game with a navigation in a virtual town, in a 15 weekly group sessions could reduce these difficulties compared to the initial assessment. This improvement could be maintained 6 months after the end of the program.
* PLANI-REV could also improve prospective memory, attention, working memory, and visuospatial organization.
* PLANI-REV could induce a clinical improvement, as well as better perception of self-efficiency, self esteem, quality of life, and conversation skills.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old.
* Diagnostic of schizophrenia or schizoaffective disorder (DSM V), attested by the MINI structured interview (Shehan et al. 1998)
* Who visit for months or year, weekly or several times per week, a day care, or therapeutic activity units outpatients clinics and nursing homes
* French Mother tongue
* Consent of the legal representative caregiver for the patients under representative law (tutelle in French).
* Clinical Stability - Therapeutic stability for at least one month.
* National healthcare assurance

Exclusion Criteria:

* Central Neurological or non stabilized somatic diseases.
* Treatments for somatic disease with putative psychotropic effect.
* Electroconvulsive therapy in the last six months
* Illetrism
* IQ< 70 established with the f-NART.
* Substance misuse or dependence (except Nicotine) or toxic for more than 5 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2024-08-09 (Estimated); Study Completion 2024-08-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PLANI-REV : questionnaire scores | 10 months
  the comparison pre/post PLANI-REV of the number of difficulties of daily life using the Profinteg questionnaire

SECONDARY OUTCOMES:
- Profinteg scores 6 months after PLANI-REV. Number of problematic activities; average score for difficulties of problematic activities. | 16 months
  To improve pre/post PLANI-REV and 6 months after, neuropsychological performances in prospective memory, attention, working memory, executive functions, and visual and spatial organization

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle AMADO, MD, Principal Investigator — CHSA
Locations (4):
- France (4):
  - Centre Hospitalier DURANT, Étampes
  - Hopital les Murets, La Queue-en-Brie
  - Centre Hospitalier Sainte Anne, Paris
  - Centre Hospitalier Guillaume Régnier, Rennes

IPD SHARING:
Plan to Share IPD: No